CLINICAL TRIAL: NCT00195234
Title: A Phase 1 Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of an HIV CTL Multi-Epitope Peptide Vaccine Formulated With RC529-SE and GM-CSF Given to HIV-1 Positive Adults on Stable HAART.
Brief Title: Study Evaluating Vaccine in Adults With HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6112K2-100
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: HIV CTL MEP 1000 micrograms, 19 months per subject

SUMMARY:
The purpose of this study is to learn whether the study vaccine and adjuvants (drugs that are used to help improve immune responses) have an acceptable safety profile in treating individuals with HIV.

A second purpose of this study is to understand how the immune system responds to the study vaccine and adjuvants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age diagnosed with HIV and on stable HAART for a minimum of six months
* CD4 T-cell count greater than and equal to 350/mm3 at screening
* No reported CD4 T-cell count less than 350/mm3 at any time before screening
* Viral load less than 50 copies/mL at screening and no viral load greater than 400 copies/mL for a minimum of six months prior to screening

Exclusion Criteria:

* Any chronic symptomatic infection other than HIV
* Use of any prior HIV vaccine (prophylactic and/or therapeutic) within one year before or during screening
* Any malignancy that may require systemic therapy
* Use of any investigational treatment within six months before screening or planned during study enrollment, except for investigational retrovirals obtained through ACTG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of the HIV CTL MEP vaccine formulated with adjuvants, administered by intramuscular (IM) injection to HIV Pos adults receiving stable HAART. Subjects will receive vaccinations at months 0, 1, 3, and 6.

SECONDARY OUTCOMES:
To evaluate the subject immune system responds to the vaccinations. To evaluate RNA and protein patterns in the collected blood samples after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (9):
- United States (9):
  - Sacramento, California
  - Denver, Colorado
  - Chicago, Illinois
  - New York, New York
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas